CLINICAL TRIAL: NCT02148575
Title: Integrating Palliative Care Into Self-Management of Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1307012400
Record Dates: First submitted 2014-05-21; First posted 2014-05-28 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2016-06

CONDITIONS: Breast Cancer
Keywords: Palliative Care; Self-management; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-Management Group (Experimental): Managing Cancer Care: A Personal Guide (MCC) is a set of magazine-format, printed modules that includes information about key self-management topics, worksheets, "conversation starters", and targeted links to local and internet resources, among other features.
  Interventions: Behavioral: Self-Management Group
- Symptom Management Group (Active Comparator): Participants in the Symptom Management Group will be given a symptom management toolkit that provides information on the most commonly experienced symptoms and side effects of cancer treatment, including fatigue, nausea, and sleep problems, among others. Each chapter includes information on when and why the symptom may occur, how the symptom can be managed, and when to call a provider.
  Interventions: Behavioral: Symptom Management Group

INTERVENTIONS:
Behavioral: Self-Management Group
  Arms: Self-Management Group
Behavioral: Symptom Management Group
  Arms: Symptom Management Group

SUMMARY:
The purpose of this study is to test a psycho-educational intervention, Managing Cancer Care: A Personal Guide (MCC), that is intended to improve patients' knowledge of palliative care and to facilitate its timely integration into self-management of their breast cancer. The MCC will be tested with patients with Stage I-IV breast cancer at baseline, one, and three months following enrollment. The intervention group will receive the MCC, and the attention-control group will receive a symptom management toolkit. Participants' family caregivers will also be enrolled to provide information on patients' self-management. Investigators hypothesize that users of MCC, as compared to attention-control participants, will demonstrate improved knowledge, feelings, and behaviors related to self-management of their cancer care. This innovative research can help to establish palliative care as a mainstay of self-management interventions that target serious illnesses.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 21
* Stage I-IV breast cancer
* Live in the State of Connecticut
* Speak English
* Receiving any kind of treatment for breast cancer
* Prognosis of at least 6 months

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2014-06; Primary Completion 2016-04 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Knowledge of Care Options Test | 1 month
Knowledge of Care Options Test | 3 months
Knowledge of Care Options Test | baseline

SECONDARY OUTCOMES:
Control Preferences Scale | 1 month
Medical Communication Competence Scale | 1 month
Measurement of Transitions Scale | 1 month
Chronic Disease Self-Efficacy Scale | 1 month
Hospital Anxiety and Depression Scale | 1 month
Uncertainty in Illness Scale | 1 month
Health Care Utilization Form | 3 months
Goals of Care Conversations Form | 1 month
Control Preferences Scale | 3 months
Medical Communication Competence Scale | 3 months
Measurement of Transitions Scale | 3 months
Chronic Disease Self-Efficacy Scale | 3 months
Hospital Anxiety and Depression Scale | 3 months
Uncertainty in Illness Scale | 3 months
Goals of Care Conversations Form | 3 months
Control Preferences Scale | baseline
Medical Communication Competence Scale | baseline
Measurement of Transitions Scale | baseline
Chronic Disease Self-Efficacy Scale | baseline
Hospital Anxiety and Depression Scale | baseline
Uncertainty in Illness Scale | baseline
Goals of Care Conversations Form | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dena Schulman-Green, PhD, Principal Investigator — Principal Investigator
Locations (2):
- United States (2):
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Yale School of Nursing, West Haven, Connecticut

REFERENCES:
- [Derived] Schulman-Green D, Linsky S, Jeon S, Kapo J, Blatt L, Chagpar A. Integrating palliative care into self-management of breast cancer: Protocol for a pilot randomized controlled trial. Contemp Clin Trials. 2016 May;48:133-8. doi: 10.1016/j.cct.2016.04.009. Epub 2016 Apr 20. PMID 27107680